CLINICAL TRIAL: NCT05500248
Title: Impact of Computer-aided Optical Diagnosis (CADx) in Predicting Histology of Diminutive Rectosigmoid Polyps: a Multicenter Prospective Trial.
Brief Title: Artificial Intelligence for Leaving in Situ Colorectal Polyps.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Giulio Antonelli, Principal Investigator, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRACTICE
Record Dates: First submitted 2022-08-11; First posted 2022-08-15 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2024-10

CONDITIONS: Colonic Neoplasms
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Leave-In-Situ Arm (Experimental): standard, high-definition colonoscopy with the use of Medtronic GI Genius module including both CADe and CADx. Polyps will be left in situ if diminutive (≤5 mm) in size, located in the rectum or sigma and optically diagnosed by the endoscopist using the system to be hyperplastic with high confidence, otherwise resected and sent to pathology.
  Interventions: Behavioral: Leave In Situ
- Standard arm (Active Comparator): standard, high-definition colonoscopy with the use of Medtronic GI Genius module including both CADe and CADx. All detected polyps regardless of size and optical diagnosis will be resected and sent to pathology.
  Interventions: Behavioral: Standard

INTERVENTIONS:
Behavioral: Leave In Situ — Polyps will be left in situ if diminutive (≤5 mm) in size, located in the rectum or sigma and optically diagnosed by the endoscopist using the system to be hyperplastic with high confidence, otherwise resected and sent to pathology.
  This behaviour is recommended by guidelines if the endoscopist is expert in optical diagnosis. In this case the endoscopists will be experts and they will also be helped by the CADx system that has shown to exceed the thresholds requested for use in clinical practice in previous trials.
  Arms: Leave-In-Situ Arm
Behavioral: Standard — All identified polyps will be removed and sent to pathology.
  Arms: Standard arm

SUMMARY:
This two parallel-arms, randomized, multicenter trial is aimed at investigating safety and effectiveness of a Computer-Aided-Diagnosis (CADx)-assisted leave-in-situ strategy (Leave-In-Situ Arm) as opposed to a resect-all strategy (Standard Arm) as implemented by endoscopists in a real-world setting.

With this study it will be possible to understand the impact of CADx in patient treatment and management both in terms of clinical outcome and costs.

DETAILED DESCRIPTION:
Real-time diminutive (≤5 mm) colonic polyp characterization by virtual blue-light (i.e. Narrow Banding Imaging [NBI], Blue Light Imaging [BLI], etc.) has been identified as a key goal for novel endoscopic advanced imaging techniques. The real-time prediction of polyps histology, especially of those located in the rectosigmoid, is clinically relevant as diminutive polyps represent the majority of polyps detected during colonoscopy and have a very low risk of harboring advanced histology (0.3%) and a negligible risk of invasive carcinoma (0%-0.08%).

Thus, as recommended by current guidelines, an optical diagnosis would allow diminutive polyps to be resected and discarded without pathological assessment (i.e. resect-and-discard strategy) or left in place without resection in the case of diminutive rectosigmoid hyperplastic polyps (i.e. leave-in-situ strategy), with an enormous cost-saving potential. In addition, the current policy for managing such hyperplastic-appearing polyps is poorly defined and variable from endoscopist to endoscopist. For instance, the European Society of Gastrointestinal Endoscopy (ESGE) recommends to leave-in-situ only diminutive polyps characterized as hyperplastic with high-confidence. However, it is currently unknown how many endoscopists actually do switch to the blue-light advanced imaging (when available) that is required for a high-confident diagnosis when assessing ≤5 mm hyperplastic-appearing lesions. More importantly, the Leave-in-situ strategy, poorly defined in a pre-AI era, has never been clinically validated, leaving uncertainty on the estimate of the possible false negatives generated by an inaccurate diagnosis6.

The availability of Computer-Aided-Diagnosis (CADx) tools, which may help endoscopists distinguish neoplastic from non-neoplastic polyps making the characterization process quicker and more objective, would be highly desirable and captivating.

A new system for CADx during white light endoscopy has been developed and integrated alongside a previously available Computer-Aided-Detection (CADe) tool (GI-Genius, Medtronic), making real-time characterization straightforward after polyp detection, and has been recently validated in a real time clinical trial, showing how this system exceeds the American Society of Gastrointestinal Endoscopy (ASGE) Criteria for clinical application of cost saving strategies (i.e. leave in situ and resect and discard), and equals the performance of expert endoscopists in optical diagnosis. However, this was a first study, monocentric and without randomization, with a small, albeit adequately powered, sample size. The need for larger trials is thus urgent to speed up the possible implementation of CADx in clinical practice.

Aim of this study is to clinically validate the new CADx tool for the implementation of a leave-in-situ strategy in a multicenter, randomized controlled trial.

ELIGIBILITY:
Inclusion criteria:

- All >18 years-old patients undergoing elective colonoscopy

Exclusion criteria:

* patients with personal history of colorectal cancer (CRC), or Inflammatory Bowel Disease (IBD).
* Patients affected with Lynch syndrome or Familiar Adenomatous Polyposis.
* patients with inadequate bowel preparation (defined as Boston Bowel Preparation Scale <2 in any colonic segment).
* patients with previous colonic resection.
* patients on antithrombotic therapy, precluding polyp resection.
* patients who were not able or refused to give informed written consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 919 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Adenoma Detection Rate (ADR) | 1 year
  the proportion of participants with at least one adenoma (per-patient analysis) in the two arms

SECONDARY OUTCOMES:
Adenoma Detection Rate (ADR) in the rectosigmoid tract. | 1 year
  the proportion of participants with at least one adenoma (per-patient analysis) in the rectosigmoid tract in the two arms.
Positive Predictive Value (PPV) | 1 year
  the proportion of clinically significant resected lesions among all resected lesions (per-polyp analysis) in the two arms

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Dei Castelli, Ariccia, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Antonelli G, Desideri F, Scarozza P, Andrisani G, Zerboni G, Furnari M, Bevilacqua N, Cossignani M, Di Fonzo M, Cereatti F, Navazzotti G, Antenucci C, Di Matteo FM, Bevivino G, Caruso A, Spadaccini M, Schiavone S, Grossi C, Rizkala T, Comberlato M, Bretthauer M, Sharma P, Von Renteln D, Rex DK, Correale L, Repici A, Mori Y, Iacopini F, Hassan C. Safety of artificial intelligence-assisted optical diagnosis for leaving colorectal polyps in situ during colonoscopy (PRACTICE): a non-inferiority, randomised controlled trial. Lancet Gastroenterol Hepatol. 2025 Oct;10(10):915-923. doi: 10.1016/S2468-1253(25)00140-2. PMID 40914178